CLINICAL TRIAL: NCT03179124
Title: Upper Extremity Function In Cerebral Palsy And Its Association With Balance And Trunk Control
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Research assistant, Gazi University
Other Study IDs: 214
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; trunk control; upper extremity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemiparetic cerebral palsy: Unilateral paresis in which upper extremities are more severely affected than lower extremities.
- Diparetic cerebral palsy: Lower extremities were more affected than upper extremities

SUMMARY:
Children with cerebral palsy (CP) have postural control problems due to the lack of motor and sensory development. Trunk control which has an important role in ensuring postural control, is the basis for sitting, mobility, development of the upper extremity, pulmonary function and activities of daily living. Poor postural control restricts upper extremity functions which also affects the quality of movements. For this reason, it is important to assess the relationship between trunk control and upper extremity functions. This study is planned to investigate the effect of balance and trunk control on upper extremity functions in children with CP.

DETAILED DESCRIPTION:
30 hemiparetic and 32 diparetic CP, in total 62 children, aged between 5-12 years, were included in this study. Trunk Control Measurement Scale (TCMS) was used to assess trunk control, Pediatric Balance Scale (PBS) was used to assess balance, and Quality of Upper Extremity Skills Test was used to assess upper extremity functions (QUEST).

ELIGIBILITY:
Inclusion Criteria:

* spastic hemiparetic and / or diparetic CP
* co-operative enough to understand test directives
* between 5 and 12 years of age
* Having spasticity of 0-2 according to the modified wax and / or modified Ashworth Scale (MAS)
* GMFCS I, II and III

Exclusion Criteria:

Have had previous orthopedic surgery to the upper extremity

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cerebral palsy (CP) describes a group of permanent disorders in movement and posture that limit activity and participation and are attributed to non-progressive disturbances in the developing fetal or infant brain
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
Quality of Upper Extremity Skills Test | 30 minutes
  QUEST is a reliable tool for children with CP aged 2-12 years.The QUEST groups upper limb movement into four domains. Each domain focuses on areas of difficulty typically seen in children with spastic cerebral palsy: (a) Dissociated Movements, (ability to voluntarily isolate movement at the shoulder, elbow, wrist and fingers); (b) Grasps (which also rates sitting postures during grasps of 1 inch cube, cereal, pencil or crayon); (c) Weight Bearing (ability to lean on the arms in prone or 4-point kneeling, sitting and while reaching); and (d) Protective Extension (using the arms to stop oneself from falling forward, backward and to the side). In addition to the four domains of movement the QUEST also has three scales: Hand Function, Spasticity and Co-operativeness.

SECONDARY OUTCOMES:
Pediatric Balance Scale | 20 minutes
  The PBS measure can be performed without specialized equipment and is quickly and easily administered. The PBS has been used to measure the balance functions for school-age children with mild-to-moderate motor impairments
Trunk Control Measurement Scale | 20 minutes
  This scale consists of 15 items measuring two main components of trunk control: (a) a stable base of support (static sitting balance), and (b) an actively moving body segment (dynamic sitting balance). The subscale static sitting balance (items 1-5) evaluates the ability of the child to maintain a stable trunk posture during movements of upper and lower limbs. The section dynamic sitting balance is further divided into two subscales: selective movement control and dynamic reaching. The subscale selective movement control (items 6-12) measures selective trunk movements in the sagittal (flexion/extension), frontal (lateral flexion) and transverse (rotation) plane within the base of support. The subscale dynamic reaching (items 13-15) evaluates the performance of three reaching tasks, requiring active trunk movements beyond the base of support

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Study Chair — study chair

IPD SHARING:
Plan to Share IPD: No